CLINICAL TRIAL: NCT06390540
Title: The Effect of Mobile-Based Exercise Application in the Postpartum Period on Depressive Symptoms, Maternal Attachment and Baby Crying: A Randomized Controlled Study
Brief Title: Mobile-Based Exercise in Postpartum Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: republic of turkey ministry of health (Unknown)
Responsible Party: Principal Investigator, Serap Canli, Public Health Nurse Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANKARA-UNALS-001
Record Dates: First submitted 2024-04-19; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Depression; Mother-Infant Interaction
Keywords: postpartum period; depression; mothers; exercise; babies and infants
MeSH Terms: conditions — Depression, Postpartum; Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This research will be conducted in accordance with the pre-test-post-test experimental research model in two groups in order to determine the effect of a mobile-based breathing and relaxation exercise program applied to postpartum women on postpartum depression, mother-infant attachment and baby crying behavior.
Who Masked: Participant
Masking Description: In the PASS 11 program, when the number of groups is calculated as 2, 5% margin of error and 90% power, it has been determined that at least 54 people should be included in the sample, with each group consisting of at least 27 people. Considering that the women taking part in the study may want to leave the study while it is ongoing and may encounter unexpected medical conditions and may be lost; It was decided to include a total of 80 women, 40 in the intervention group and 40 in the control group. In this single-blind randomized controlled study, the group in which women will be included will be determined and randomized via computer. "Random Allocation Software Program" will be used to randomize women to groups. The randomization process will be generated by the computer into random blocks of permuted length. Women will be assigned to one of the intervention and control groups by the researchers according to the order in the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): In the study, women will perform breathing and relaxation exercises for 8 weeks.
  In the first phase of the intervention, women will be given home exercise program training. The training will be held face to face at the Family Health Center. The day and time will be determined according to the women's preference. Afterwards, women will be informed about the exercise program and the exercise program will be shared in writing.
  In the second phase of the intervention, a total of four exercise videos will be sent to women every two weeks on Sunday.Exercise videos will be sent to women through social networks such as WhatsApp, Instagram, Facebook and Twitter.
  Women's exercise routines will be recorded by researchers by calling the women and monitoring whether they do the exercises through self-report.
  Interventions: Other: Exercise
- Control Group (No Intervention): No intervention will be made to women in the control group. When necessary, women's questions will be answered via phone. At the end of the study, breathing and relaxation exercise training will be given to the control group. Trainings will be held face to face at the Family Health Center. The training program will be planned taking into account the demands of women.

INTERVENTIONS:
Other: Exercise — During the training, verbal information will be given about the importance of exercise, exercise barriers, and the potential benefits of exercise on the mother and baby in the postpartum period. In the training, the points that the mother should pay attention to before exercise will also be discussed. In the following process, videos containing deep breathing and relaxation exercises will be sent to women. The videos will be recorded by the researchers at Ankara University Physiotherapy application laboratory. Recording videos will be delivered to women through social networks. Women will be allowed to do these exercises for a total of 8 weeks.
  Arms: Exercise Group

SUMMARY:
Postpartum depression is a global mental health problem affecting 13 million women worldwide each year. It is defined as minor or major depression that occurs up to one year after birth and is estimated to affect 5 to 25% of mothers who have just given birth . Postpartum depression can cause negative consequences not only on the mother but also on the newborn and the whole family. The main goal in the postpartum period is to maintain the well-being of mother and baby. However, if a depression is experienced during this period, the main goal is to take action to reduce its severity. Exercise is a potentially promising method to prevent postpartum depression. However, more studies are needed to determine the effects of exercise on women who live in rural Türkiye and have limited access to health services. Therefore, this study aims to determine the effect of a mobile-based exercise program applied to women giving birth in rural areas on postpartum depression, mother-baby attachment and baby crying behavior.

DETAILED DESCRIPTION:
Postpartum depression is a global mental health problem affecting 13 million women worldwide each year . It is defined as minor or major depression that occurs up to one year after birth and is estimated to affect 5 to 25% of mothers who have just given birth . Postpartum depression, often associated with periodic depressive episodes, is characterized by emotional lability, guilt, dysphoria, disorientation, and suicidal thoughts and can persist for a long time. Postpartum depression is recognized as an official diagnosis by the World Health Organization's International Classification of Disorders, 10th revision (ICD-10) and the Diagnostic and Statistical Manual of Mental Disorders. While ICD-10 reports that the most critical period for diagnosing postpartum depression is within six weeks after birth, the American Psychiatric Association reported that episodes of postpartum depression can begin within four weeks after birth. Postpartum depression can also turn into permanent and long-term depression, which can increase the likelihood of recurrent episodes of depression in subsequent pregnancies. This is supported by evidence that women with a history of depressive illness are more likely to develop postpartum depression. Postpartum depression can cause negative consequences not only on the mother but also on the newborn and the whole family. Postpartum depression, in particular, has significant effects on mother-infant attachment; It also has negative effects on the mother learning how to care for her baby and transitioning into the parenting role. Postpartum depression can lead to early cessation of breastfeeding or breastfeeding problems; It may also cause the use of preventive health services and vaccination rates in children to be low. Impairments in social participation and emotional regulation, increased negative emotionality, and high cortisol reactivity may be observed in babies of mothers with depression.

During the postpartum period, not only mothers but also their babies may show some behavioral reactions. One of these is crying. There are many possible causes of crying problems in babies, but none of them are certain. It has generally focused on conditions that cause excessive crying in the baby, such as immaturity of the intestinal flora, cow's milk allergy and intestinal microbiota composition. Many studies have raised the question of whether the cause may lie in maternal factors. Crying problems in babies have been associated with low maternal age and education level. Some researchers agree that crying problems arise from the complex mother-infant dyad, and it is well known that maternal postpartum depression and infant crying influence each other . Systematic reviews on this topic have generally found associations between the mother's mental problems (stress, anxiety, or depression) during pregnancy and the baby's regulatory problems, including crying.

The main goal in the postpartum period is to maintain the well-being of mother and baby. However, if a depression is experienced during this period, the main goal is to take action to reduce its severity. Postpartum depression is a specific psychological disorder for which preventive interventions can provide dramatic benefits. In their meta-analysis study by It has been stated that practices such as cognitive behavioral therapies, social support groups, psycho-educational training, physical exercises, yoga, and lack of nutritional supplements are interventions that can be used to reduce the severity of postpartum depression..

Exercise is a potentially promising method to prevent postpartum depression. Since the aim of exercise is to improve or maintain one or more aspects of physical fitness, it is defined as a planned, systematic, repeated and purposeful action.Previous studies have provided compelling evidence regarding exercise in the postpartum period. It has been reported that exercises performed in the postpartum period provide psychosocial well-being, less anxiety and depression, better cardiovascular adaptation, body fat/weight control, less bone loss due to breastfeeding and less stress incontinence, and strengthen the bonding between mother and baby.

Studies generally point to the importance of regular exercise in the postpartum period. However, the number of women exercising in the postpartum period is limited, and lack of access to affordable and appropriate activities is a perceived barrier to exercise. The increasing number of mobile-based applications in recent years offers affordable and accessible exercise applications. These apps use a variety of features, from tracking exercise activity to providing motivational messages. However, what is known about whether exercise practices improve health outcomes and, if so, the mechanisms of these effects is limited. Therefore, there is a need for more studies in this important area to determine the effects of exercise using new technologies as an alternative to face-to-face exercise programs, especially for women living in rural Türkiye and with limited access to health services.

Women who give birth in Türkiye are followed up in the hospital for 24 hours and then followed up three times during the postpartum period at home or in Family Health Centers (FHC) within the scope of health services. Health professionals have a unique duty to follow up women in the postpartum period, identify women at risk for depression, and encourage mothers to use preventive practices such as exercise. It is very important for midwives and nurses to explain mobile-based exercise programs to prevent the development of depression, especially to women living in rural areas, in the postpartum period, to persuade women to participate in these programs, and to perform exercises regularly under the supervision of doctors and physiotherapists in terms of protecting the health of women and their families. Therefore, the aim of this study is to determine the effect of a mobile-based exercise program applied to women giving birth in rural areas on reducing the severity of postpartum depression, mother-baby bonding, and baby crying behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Having had a singleton pregnancy,
2. Not having a history of serious illness/chronic disease,
3. Not being restricted from exercising by the physician,
4. Having given birth at term (37-42 weeks of pregnancy),
5. Being within the first 6 months after birth,
6. Having a healthy baby,
7. Knowing how to read and write Turkish and understanding it,
8. Having the skills to use phones, tablets, computers and mobile applications,
9. Not having any problems that would prevent communication,
10. Agreeing to participate in the research. -

Exclusion Criteria:

1. Having a history of multiple pregnancy,
2. Being taking medication for the treatment of illness or chronic disease,
3. Exercising regularly,
4. Having a premature baby (<37 weeks of gestation),
5. Having a history of illness in the baby,
6. Not having a phone, tablet or computer,
7. Not agreeing to participate in the research. -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility of participants is based on female gender representation.
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Chance from Baseline in Depression on the 30-point Edinburgh Postpartum Depression Scale at Week 8 | Baseline and 8 week
  The Edinburgh Postpartum Depression Scale is a validated, self-reported instrument assessing average depression intensify postpartum period. Possible scores range from 0 (no depression) to 30 (depression).
  The scale consists of 10 questions in total. Each question provides a four-point Likert type measurement. The items in questions 3, 5, 6, 7, 8, 9 and 10 of the scale are scored as 3, 2, 1, 0 and gradually indicates decreasing intensity. The scoring of the items in questions 1, 2 and 4 is in the form of 0, 1, 2, 3, indicating increasing severity. By summing these items, the total score of the scale is obtained. The lowest total score that can be obtained on the scale is 0 and the highest is 30.

SECONDARY OUTCOMES:
Chance from Baseline in Mother-baby attachment on the 104-point Maternal Attachment Scale at Week 8 | Baseline and 8 week
  The Maternal Attachment Scale is a validated, self-reported instrument assessing average attachment with maternal love. Possible scores range from 26 (low attachment) to 104 (high attachment).
  The Maternal Attachment scale is a 4-point Likert type scale with 26 questions. The items in the scale consist of the options "never-1 point", "sometimes-2 points", "often-3 points", "always-4 points". Each item in the scale consists of a positive structure and is scored. The maximum score that women can get from the scale is "104" and the minimum score is "26". The highest score obtained from the scale is maternal in women. The lowest score indicates that maternal attachment is low in women.

OTHER OUTCOMES:
Chance from Baseline in baby criying Baby Cry Diary at Week 8 | Baseline and 8 week
  The Infant Cry Diary is a self-reported tool that assesses infant crying over a 24-hour period.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu YM, McArthur E, Dixon S, Dirk JS, Welk BK. Association between intrapartum epidural use and maternal postpartum depression presenting for medical care: a population-based, matched cohort study. Int J Obstet Anesth. 2018 Aug;35:10-16. doi: 10.1016/j.ijoa.2018.04.005. Epub 2018 Apr 21. PMID 29954649
- [Background] Tonei V. Mother's mental health after childbirth: Does the delivery method matter? J Health Econ. 2019 Jan;63:182-196. doi: 10.1016/j.jhealeco.2018.11.006. Epub 2018 Dec 7. PMID 30594609
- [Background] Zhou C, Hu H, Wang C, Zhu Z, Feng G, Xue J, Yang Z. The effectiveness of mHealth interventions on postpartum depression: A systematic review and meta-analysis. J Telemed Telecare. 2022 Feb;28(2):83-95. doi: 10.1177/1357633X20917816. Epub 2020 Apr 19. PMID 32306847
- [Background] Carter T, Bastounis A, Guo B, Jane Morrell C. The effectiveness of exercise-based interventions for preventing or treating postpartum depression: a systematic review and meta-analysis. Arch Womens Ment Health. 2019 Feb;22(1):37-53. doi: 10.1007/s00737-018-0869-3. Epub 2018 Jun 7. PMID 29882074
- [Background] Saligheh M, McNamara B, Rooney R. Perceived barriers and enablers of physical activity in postpartum women: a qualitative approach. BMC Pregnancy Childbirth. 2016 Jun 2;16(1):131. doi: 10.1186/s12884-016-0908-x. PMID 27256279
- [Background] Payne JL, Maguire J. Pathophysiological mechanisms implicated in postpartum depression. Front Neuroendocrinol. 2019 Jan;52:165-180. doi: 10.1016/j.yfrne.2018.12.001. Epub 2018 Dec 12. PMID 30552910
- [Background] Hoifodt RS, Nordahl D, Pfuhl G, Landsem IP, Thimm JC, Ilstad LKK, Wang CEA. Protocol for the Northern babies longitudinal study: predicting postpartum depression and improving parent-infant interaction with The Newborn Behavioral Observation. BMJ Open. 2017 Sep 27;7(9):e016005. doi: 10.1136/bmjopen-2017-016005. PMID 28963284
- [Background] Kasamatsu H, Tsuchida A, Matsumura K, Shimao M, Hamazaki K, Inadera H; Japan Environment and Children's Study Group. Understanding the relationship between postpartum depression one month and six months after delivery and mother-infant bonding failure one-year after birth: results from the Japan Environment and Children's study (JECS). Psychol Med. 2020 Jan;50(1):161-169. doi: 10.1017/S0033291719002101. Epub 2019 Sep 2. PMID 31474232
- [Background] Reijneveld SA, Brugman E, Hirasing RA. Excessive infant crying: the impact of varying definitions. Pediatrics. 2001 Oct;108(4):893-7. doi: 10.1542/peds.108.4.893. PMID 11581441
- [Background] Cirgin Ellett ML. What is known about infant colic? Gastroenterol Nurs. 2003 Mar-Apr;26(2):60-5. doi: 10.1097/00001610-200303000-00004. PMID 12682526
- [Background] Loughman A, Quinn T, Nation ML, Reichelt A, Moore RJ, Van TTH, Sung V, Tang MLK. Infant microbiota in colic: predictive associations with problem crying and subsequent child behavior. J Dev Orig Health Dis. 2021 Apr;12(2):260-270. doi: 10.1017/S2040174420000227. Epub 2020 Apr 13. PMID 32279681
- [Background] Petzoldt J, Wittchen HU, Einsle F, Martini J. Maternal anxiety versus depressive disorders: specific relations to infants' crying, feeding and sleeping problems. Child Care Health Dev. 2016 Mar;42(2):231-45. doi: 10.1111/cch.12292. Epub 2015 Oct 22. PMID 26490836
- [Background] Papousek M, von Hofacker N. Persistent crying in early infancy: a non-trivial condition of risk for the developing mother-infant relationship. Child Care Health Dev. 1998 Sep;24(5):395-424. doi: 10.1046/j.1365-2214.2002.00091.x. PMID 9728285
- [Background] Raiha H, Lehtonen L, Huhtala V, Saleva K, Korvenranta H. Excessively crying infant in the family: mother-infant, father-infant and mother-father interaction. Child Care Health Dev. 2002 Sep;28(5):419-29. doi: 10.1046/j.1365-2214.2002.00292.x. PMID 12296876
- [Background] Olmestig TK, Siersma V, Birkmose AR, Kragstrup J, Ertmann RK. Infant crying problems related to maternal depressive and anxiety symptoms during pregnancy: a prospective cohort study. BMC Pregnancy Childbirth. 2021 Nov 17;21(1):777. doi: 10.1186/s12884-021-04252-z. PMID 34789174
- [Background] Petzoldt J. Systematic review on maternal depression versus anxiety in relation to excessive infant crying: it is all about the timing. Arch Womens Ment Health. 2018 Feb;21(1):15-30. doi: 10.1007/s00737-017-0771-4. Epub 2017 Sep 13. PMID 28900745
- [Background] Korja R, Nolvi S, Grant KA, McMahon C. The Relations Between Maternal Prenatal Anxiety or Stress and Child's Early Negative Reactivity or Self-Regulation: A Systematic Review. Child Psychiatry Hum Dev. 2017 Dec;48(6):851-869. doi: 10.1007/s10578-017-0709-0. PMID 28124273
- [Background] Caparros-Gonzalez RA, Torre-Luque A, Romero-Gonzalez B, Quesada-Soto JM, Alderdice F, Peralta-Ramirez MI. Stress During Pregnancy and the Development of Diseases in the offspring: A Systematic-Review and Meta-Analysis. Midwifery. 2021 Jun;97:102939. doi: 10.1016/j.midw.2021.102939. Epub 2021 Feb 23. PMID 33647755
- [Background] Reck C, Tietz A, Muller M, Seibold K, Tronick E. The impact of maternal anxiety disorder on mother-infant interaction in the postpartum period. PLoS One. 2018 May 25;13(5):e0194763. doi: 10.1371/journal.pone.0194763. eCollection 2018. PMID 29799842
- [Background] Santona A, Tagini A, Sarracino D, De Carli P, Pace CS, Parolin L, Terrone G. Maternal depression and attachment: the evaluation of mother-child interactions during feeding practice. Front Psychol. 2015 Aug 24;6:1235. doi: 10.3389/fpsyg.2015.01235. eCollection 2015. PMID 26379576
- [Background] Brockington IF, Aucamp HM, Fraser C. Severe disorders of the mother-infant relationship: definitions and frequency. Arch Womens Ment Health. 2006 Sep;9(5):243-51. doi: 10.1007/s00737-006-0133-0. Epub 2006 May 15. PMID 16699838
- [Background] Sockol LE, Epperson CN, Barber JP. Preventing postpartum depression: a meta-analytic review. Clin Psychol Rev. 2013 Dec;33(8):1205-17. doi: 10.1016/j.cpr.2013.10.004. Epub 2013 Oct 21. PMID 24211712
- [Background] Dasso NA. How is exercise different from physical activity? A concept analysis. Nurs Forum. 2019 Jan;54(1):45-52. doi: 10.1111/nuf.12296. Epub 2018 Oct 17. PMID 30332516
- [Background] Larson-Meyer DE. Effect of postpartum exercise on mothers and their offspring: a review of the literature. Obes Res. 2002 Aug;10(8):841-53. doi: 10.1038/oby.2002.114. PMID 12181395
- [Background] McCurdy AP, Boule NG, Sivak A, Davenport MH. Effects of Exercise on Mild-to-Moderate Depressive Symptoms in the Postpartum Period: A Meta-analysis. Obstet Gynecol. 2017 Jun;129(6):1087-1097. doi: 10.1097/AOG.0000000000002053. PMID 28486363
- [Background] Litman L, Rosen Z, Spierer D, Weinberger-Litman S, Goldschein A, Robinson J. Mobile Exercise Apps and Increased Leisure Time Exercise Activity: A Moderated Mediation Analysis of the Role of Self-Efficacy and Barriers. J Med Internet Res. 2015 Aug 14;17(8):e195. doi: 10.2196/jmir.4142. PMID 26276227
- [Background] Ko YL, Yang CL, Chiang LC. Effects of postpartum exercise program on fatigue and depression during "doing-the-month" period. J Nurs Res. 2008 Sep;16(3):177-86. doi: 10.1097/01.jnr.0000387304.88998.0b. PMID 18792887
- [Background] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880
- [Background] Poyatos-Leon R, Garcia-Hermoso A, Sanabria-Martinez G, Alvarez-Bueno C, Cavero-Redondo I, Martinez-Vizcaino V. Effects of exercise-based interventions on postpartum depression: A meta-analysis of randomized controlled trials. Birth. 2017 Sep;44(3):200-208. doi: 10.1111/birt.12294. Epub 2017 Jun 6. PMID 28589648
- [Background] Forsyth J, Boath E, Henshaw C, Brown H. Exercise as an adjunct treatment for postpartum depression for women living in an inner city-A pilot study. Health Care Women Int. 2017 Jun;38(6):635-639. doi: 10.1080/07399332.2017.1295049. Epub 2017 Feb 14. PMID 28278021
- [Background] Mohd Shukri NH, Wells J, Eaton S, Mukhtar F, Petelin A, Jenko-Praznikar Z, Fewtrell M. Randomized controlled trial investigating the effects of a breastfeeding relaxation intervention on maternal psychological state, breast milk outcomes, and infant behavior and growth. Am J Clin Nutr. 2019 Jul 1;110(1):121-130. doi: 10.1093/ajcn/nqz033. PMID 31161202
- [Background] Coll CVN, Domingues MR, Stein A, da Silva BGC, Bassani DG, Hartwig FP, da Silva ICM, da Silveira MF, da Silva SG, Bertoldi AD. Efficacy of Regular Exercise During Pregnancy on the Prevention of Postpartum Depression: The PAMELA Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e186861. doi: 10.1001/jamanetworkopen.2018.6861. PMID 30646198
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Muller ME. A questionnaire to measure mother-to-infant attachment. J Nurs Meas. 1994 Winter;2(2):129-41. PMID 7780768
- [Background] McRury JM, Zolotor AJ. A randomized, controlled trial of a behavioral intervention to reduce crying among infants. J Am Board Fam Med. 2010 May-Jun;23(3):315-22. doi: 10.3122/jabfm.2010.03.090142. PMID 20453177
- [Background] Baljon KJ, Romli MH, Ismail AH, Khuan L, Chew BH. Effectiveness of breathing exercises, foot reflexology and back massage (BRM) on labour pain, anxiety, duration, satisfaction, stress hormones and newborn outcomes among primigravidae during the first stage of labour in Saudi Arabia: a study protocol for a randomised controlled trial. BMJ Open. 2020 Jun 15;10(6):e033844. doi: 10.1136/bmjopen-2019-033844. PMID 32540887
- [Background] Liu X, Wang G, Cao Y. Physical exercise interventions for perinatal depression symptoms in women: A systematic review and meta-analysis. Front Psychol. 2022 Dec 13;13:1022402. doi: 10.3389/fpsyg.2022.1022402. eCollection 2022. PMID 36582320
- [Background] ACOG Committee Obstetric Practice. ACOG Committee opinion. Number 267, January 2002: exercise during pregnancy and the postpartum period. Obstet Gynecol. 2002 Jan;99(1):171-3. doi: 10.1016/s0029-7844(01)01749-5. PMID 11777528
- [Background] Aydin N, Inandi T, Yigit A, Hodoglugil NN. Validation of the Turkish version of the Edinburgh Postnatal Depression Scale among women within their first postpartum year. Soc Psychiatry Psychiatr Epidemiol. 2004 Jun;39(6):483-6. doi: 10.1007/s00127-004-0770-4. PMID 15205733
- See also: NCSS. User's Guide I Quick Start, Proportions, and Diagnostic Tests PASS Power Analysis and Sample Size System — http://www.ncss.com/wp-content/uploads/2012/09/PASS11UG1.pdf
- See also: T.C. Haymana Kaymakamlığı — http://www.haymana.gov.tr/ilcemiz-nufusu